CLINICAL TRIAL: NCT02330887
Title: Group Antenatal Care: The Power of Peers for Increasing Skilled Birth Attendance in Achham, Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Possible (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GroupANCnyaya
Record Dates: First submitted 2014-12-31; First posted 2015-01-05 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Prenatal Care
Keywords: Maternal Mortality; Institutional Birth Rate; Neonatal Mortality Rate; Preterm Birth; Stillbirth; Infant, Small for Gestational Age; Nepal; Implementation Research; Global Health
MeSH Terms: conditions — Maternal Death; Premature Birth; Stillbirth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Cohort (Experimental): We will use a cohort of 60 women from intervention village clusters for the group antenatal care intervention.
  Interventions: Other: Group Antenatal Care
- Control Cohort (Active Comparator): We will use a cohort of 60 women from control village clusters as an active comparison.
  Interventions: Other: Individual Antenatal Care

INTERVENTIONS:
Other: Group Antenatal Care — The group antenatal care intervention will match pregnant women by gestational age in the intervention village clusters and assign them to peer group sessions facilitated by local healthcare clinic staff.
  Arms: Intervention Cohort
Other: Individual Antenatal Care — Pregnant women in control village clusters will have individual antenatal care sessions with their healthcare provider.
  Arms: Control Cohort

SUMMARY:
In rural Nepal, the major drivers of underutilization of skilled birth attendance are poverty, poor social support and inadequate birth planning. Drawing from similar programs that have been shown to improve maternal and neonatal outcomes, we have designed a group antenatal care program that uses a participatory learning and action process to engage women in identifying and solving problems accessing maternity care services and create a supportive social network. We plan to test a group antenatal care program that will change antenatal care in three major ways: 1) conduct care in a group setting with women matched by gestational age, 2) incorporate participatory learning and action, and 3) provide expert and facilitated peer counseling.

DETAILED DESCRIPTION:
The group antenatal care intervention aims to improve rates of institutional birth and ANC care completion via improving acceptability of group care, maternal and neonatal health knowledge, self-efficacy, social support, and birth planning.

Objective 1: Assess the effect of group antenatal care on institutional birth rates through a prospective study using community household census data. Secondary outcomes will be completion of basic ANC package; neonatal mortality rate; percentage of preterm births; percentage of stillbirths; and percentage of small-for-gestational age (SGA) births.

* Hypothesis 1: Group ANC will increase institutional birth rates by 5% over one year.
* Hypothesis 2: Group ANC will increase completion of 4 ANC visits by 5% over one year.
* Hypothesis 3: Group ANC will reduce infant mortality rate by 5% over one year.
* Hypothesis 4: Group ANC will reduce the postpartum contraceptive prevalence rate by 5% over one year.
* Hypothesis 5: Group ANC will reduce the stillbirth rate by 5% over one year.
* Hypothesis 6: Group ANC will reduce the perinatal mortality rate 5% over one year.
* Hypothesis 7: Group ANC will reduce the combined infant mortality and stillbirth rate by 5% over one year.

Objective 2: Assess the mechanisms of implementation of group antenatal care through quantitative participant survey measures, qualitative focus group discussions and key informant interviews.

* Hypothesis 1: Group antenatal care will be acceptable to participants and providers, and preferred to individual care.
* Hypothesis 2: Group antenatal care will increase pregnant patients' access to and utilization of delivery services through improved knowledge, self-efficacy, social support and birth planning.

Objective 3: Report on key aspects of the implementation process: costs, human resources, logistics, and fidelity of the group antenatal program to model content and participatory processes.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 15-49 years old
* Resident of 14 village clusters in study site
* Intervention cohort: less than 24 weeks' gestation prior to first group antenatal care session.

Exclusion Criteria:

* Intervention cohort: more than 24 weeks' gestation prior to first group antenatal care session.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2184 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-07-10 (Actual); Study Completion 2016-07-10 (Actual)

PRIMARY OUTCOMES:
Institutional Birth Rate | 1 year
  We expect the number of pregnant women from intervention village clusters who give birth at a healthcare facility to increase by 5% compared to control.

SECONDARY OUTCOMES:
Infant Mortality Rate | 1 year
  We expect the infant mortality rate to be 5% lower among the babies from the intervention cohort women compared to control.
Postpartum contraceptive prevalence rates | 1 year
  We expect the postpartum contraceptive prevalence rate to be 5% higher among the intervention cohort women compared to control.
Completion percentage of 4 antenatal care visits | 1 year
  We expect that 5% more women in the intervention cohort will complete all 4 antenatal care visits compared to the control.
Stillbirth rate | 1 year
  We expect that the stillbirth rate will be 5% lower among the intervention cohort compared to control.
Perinatal mortality rate | 1 year
  We expect that the perinatal mortality rate will be 5% lower among the intervention cohort compared to control.
Combined infant mortality and stillbirth rate | 1 year
  We expect that the combined infant mortality and stillbirth rate will be 5% lower among the intervention cohort compared to control

CONTACTS AND LOCATIONS:
Overall Officials: David Citrin, PhD, MPH, Study Director — Possible; Duncan Maru, MD, PhD, Principal Investigator — Possible; Biraj Karmacharya, MBBS, Msc, Study Chair — University of Washington
Locations (1):
- Bayalpata Hospital, Bayaplata, Achham, Nepal

REFERENCES:
- [Derived] Harsha Bangura A, Nirola I, Thapa P, Citrin D, Belbase B, Bogati B, B K N, Khadka S, Kunwar L, Halliday S, Choudhury N, Schwarz R, Adhikari M, Kalaunee SP, Rising S, Maru D, Maru S. Measuring fidelity, feasibility, costs: an implementation evaluation of a cluster-controlled trial of group antenatal care in rural Nepal. Reprod Health. 2020 Jan 17;17(1):5. doi: 10.1186/s12978-019-0840-4. PMID 31952543
- [Derived] Thapa P, Bangura AH, Nirola I, Citrin D, Belbase B, Bogati B, Nirmala BK, Khadka S, Kunwar L, Halliday S, Choudhury N, Ozonoff A, Tenpa J, Schwarz R, Adhikari M, Kalaunee SP, Rising S, Maru D, Maru S. The power of peers: an effectiveness evaluation of a cluster-controlled trial of group antenatal care in rural Nepal. Reprod Health. 2019 Oct 22;16(1):150. doi: 10.1186/s12978-019-0820-8. PMID 31640770
- See also: Possible — http://possiblehealth.org/
- See also: Healthcare Systems Design Group — http://hsdg.partners.org/